CLINICAL TRIAL: NCT04929288
Title: Sex Differences in Risk for Alcohol Use Disorder: Neural and Hormonal Influences
Brief Title: Neural and Hormonal Influences on Sex Differences in Risk for AUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica Weafer (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Jessica Weafer, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 58758; R01AA028503 (NIH)
Record Dates: First submitted 2020-11-11; First posted 2021-06-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder
Keywords: sex; inhibitory control; risk factor; hormone; fMRI; menstrual cycle
MeSH Terms: conditions — Alcoholism; Coitus | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Males (Experimental): Participants in this group will be adult male drinkers.
  Interventions: Drug: Alcohol
- Females (Experimental): Participants in this group will be adult female drinkers. Data will be segregated by menstrual cycle phase.
  Interventions: Drug: Alcohol

INTERVENTIONS:
Drug: Alcohol — Participants will complete three experimental sessions. In each session, participants will provide detailed reports of their alcohol consumption over the past five days, and they will provide a blood sample for hormone assays. They will perform tasks during fMRI to assess each of the neurofunctional addiction domains: inhibitory control, negative emotionality, and cue reactivity. Following the fMRI scan, subjects will self-administer intravenous alcohol to provide a controlled assessment of pharmacologically-driven alcohol consumption.

SUMMARY:
The sex gap in alcohol consumption is closing rapidly, due to alarming increases among women. From 2002-2013, Alcohol Use Disorder (AUD) increased 84% for women, compared to 35% for men. As such, there is an urgent need to determine the factors underlying sex differences in risk for AUD. Current addiction models propose three domains that drive problematic alcohol use and serve as candidate sex-specific risk factors: executive function, negative emotionality, and incentive salience. Data suggest that poor inhibitory control, a key component of executive function, is a stronger risk factor for women than for men. Moreover, there is have preliminary evidence that female drinkers show less engagement of neural inhibitory circuitry, and that this sex difference is influenced by estradiol. However, the degree to which hormonally-moderated sex differences in executive function extend to the negative emotionality and incentive salience domains, and how these sex differences influence current and future drinking is unknown.

The goal of this study is to identify the mechanisms underlying sex-specific risk for AUD, and ultimately to help develop sex-specific prevention and treatment efforts. The overall objective of this trial is to determine the neural and hormonal factors contributing to sex-specific risk for AUD in three addiction domains: inhibitory control (executive function), negative emotionality, and alcohol cue reactivity (incentive salience).

ELIGIBILITY:
Inclusion Criteria:

* consume 4/5 drinks per week
* fluent in English
* high school education
* right-handed
* regular menstrual cycles (women)

Exclusion Criteria:

* serious medical problems
* body weight <110 or >210 lbs
* current medical or psychiatric conditions requiring medication for which alcohol is contraindicated
* substance use disorder other than alcohol
* current or recent history of inpatient/intensive treatment for addictive behaviors
* pregnant, nursing, on hormonal contraception
* contraindications for fMRI
* smoking > 5 cigarettes per day

Ages: 21 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Neural inhibitory function | 13 minutes
  One measure of neural inhibitory function during performance of the stop signal task will be activity (as measured by BOLD % signal change)
Neural inhibitory function | 13 minutes
  The other measure of neural inhibitory function during performance of the stop signal task will be functional connectivity for the StopInh>Go contrast.
Neural negative emotionality | 14 minutes
  One measure of neural negative emotionality during performance of the Emotional Pictures Task will be activity (as measured by BOLD % signal change)
Neural negative emotionality | 14 minutes
  The other measure of neural negative emotionality during performance of the Emotional Pictures Task will be functional connectivity for the Negative>Neutral contrast.
Neural alcohol cue reactivity | 12 minutes
  One measure of neural alcohol cue reactivity during performance of the Alcohol Cue Reactivity Task will be activity (as measured by BOLD % signal change)
Neural alcohol cue reactivity | 12 minutes
  The other measure of neural alcohol cue reactivity during performance of the Alcohol Cue Reactivity Task will be functional connectivity for the Alcohol>Neutral contrast.
Intravenous alcohol self-administration (IV-ASA) | 60 minutes
  One measure of IV-ASA will be peak BrAC (mg%; highest BrAC obtained during the IV-ASA period)
Intravenous alcohol self-administration (IV-ASA) | 60 minutes
  Another measure of IV-ASA will be whether or not a participant reached binge level of alcohol exposure (80mg%)
Intravenous alcohol self-administration (IV-ASA) | 60 minutes
  The final measure of IV-ASA will be time to reach binge level of alcohol exposure (80mg%)
Self-reported current alcohol consumption | 20 minutes
  One measure of current alcohol consumption will be number of binge days (4/5 or more drinks in a sitting for women/men) as determined by responses on the Timeline Followback.
Self-reported current alcohol consumption | 20 minutes
  The other measure of current alcohol consumption will be average peak BrAC obtained on drinking days over the past 5 days, as determined by responses on the Timeline Followback.
Prospective alcohol consumption | 18 months
  One measure of prospective alcohol consumption will be number of binge episodes as determined by responses on the 90-day Timeline Followback.
Prospective alcohol consumption | 18 months
  The other measure of prospective alcohol consumption will be drinking days per month, as determined by responses on the 90-day Timeline Followback.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Weafer, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No